CLINICAL TRIAL: NCT01176149
Title: Role Of Self-monitoring of Blood Glucose and Intensive Education in Patients With Type 2 Diabetes Not Receiving Insulin: a Pilot Study
Brief Title: Role Of Self-monitoring of Blood Glucose and Intensive Education in Patients With Type 2 Diabetes Not Receiving Insulin
Acronym: ROSES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Consorzio Mario Negri Sud (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Antonio Nicolucci / Scientific responsible, Consorzio Mario Negri Sud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSES-01
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Self monitoring blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMBG + intensive education (Experimental): Patients will receive specific educational interventions to teach them how to perform Self monitoring Blood Glucose (SMBG), how to modify diet and level of physical activity according to blood glucose levels, and the actions to be undertaken in case of abnormal values (hypoglycemia, particularly elevated glucose levels). Patients will be instructed to modify their lifestyle habits (diet, physical activity) in order to reach specific goals (weight reduction, reduction in fat consumption intake, reduction in saturated fat intake, increase in fiber intake, regular physical activity.
  Interventions: Behavioral: SMBG plus intensive education
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: SMBG plus intensive education
  Arms: SMBG + intensive education

SUMMARY:
The aim of this pilot study is to evaluate the validity and feasibility of an educational approach involving nurses, combined with SMBG, aimed at lifestyle modification and timely changes in therapy, when needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes (known diabetes or new diagnosis) seen for the first time in the diabetes outpatient clinic;
* Patients on treatment with OHA monotherapy (i.e. metformin alone or sulphonylureas alone or TZDs alone);
* No need for insulin treatment;
* Male and female patients, aged between 45-75 years;
* Hba1c values between 7% and 9% included (considering a value of 6.0% as the upper limit of normal value)
* No experience of self monitoring of blood glucose in the previous 12 months (SMBG performed with a frequency of < 1 times/week)
* Ability and willingness to comply with all study requirements
* Signature of consent form

Exclusion Criteria:

* Patients incapable to perform SMBG
* Patients needing insulin or multiple OHA association therapy
* Patients needing a regular use of SMBG (e.g. frequent hypoglycemic episodes)
* Diabetes care not exclusively managed by diabetic clinics
* Patients with serious underlying medical or psychiatric condition

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Improvement of metabolic control
  Aim of this study is to evaluate the efficacy of Self Monitoring Blood Glucose and Intensive Education in terms of improvement of metabolic control expressed as HbA1c levels after 6 months.

SECONDARY OUTCOMES:
Reduction in prandial Blood Glucose excursions
Percentage of patients needing therapy modifications
Percentage of patients reaching target HbA1c (i.e. <7.0%)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nicolucci, MD, Study Director — Consorzio Mario Negri Sud
Locations (1):
- Consorzio Mario Negri Sud, Santa Maria Imbaro, Chieti, Italy